CLINICAL TRIAL: NCT05606679
Title: Maternal KIR and Fetal HLA Influence Reproductive Success in ART-oocyte Donor.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IVI Madrid (Other)
Collaborators: Diana Alecsandru (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2207-MAD-098-DA
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Reproductive Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing ART with oocyte donation: Healthy patients with no history of RIF and RM which have undergone or are undergoing ART with oocyte donation and SET.
  Interventions: Genetic: Analysis combinations of maternal KIR and HLA-C genotypes

INTERVENTIONS:
Genetic: Analysis combinations of maternal KIR and HLA-C genotypes — Analysis of combinations of maternal KIR and HLA-C genotypes of the egg donor and fetus (based on the genotypes of the donor and male partner), as well as different HLA-F SNP genotypes of the recipients

SUMMARY:
The present project is an ambispective study designed to answer how HLA-F SNPs, as well as KIR-HLA-C compatibility, influence reproductive outcomes in oocyte donation cycles. On the one hand, healthy patients without history of RIF and RM and with indication of egg donation cycle as ART treatment will be genotype for KIR, HLA-C and HLA-F. HLA-C from male partners and egg donors will be also analyzed. No matching based on HLA-C genotypes would be performed and donors would be assigned to recipients following the routine clinical practices. After SET, patients will be followed up until delivery or until the end of treatment. On the other hand, access to data from patients who have equally undergone oocyte-donation cycles, who meet the inclusion criteria and who have been genotyped for KIR and HLA-C as a matter of routine practice, will be requested.

For this study, only the first SET of oocyte-donation that patients undergo will be considered. LBR will be the primary endpoint of the study. In addition, secondary endpoints such as embryo development, sustained implantation, progesterone levels, implantation failure, miscarriage rate and unwanted events (preeclampsia, fetal grow restriction, premature birth, low birth weight…) will also be evaluated.

DETAILED DESCRIPTION:
This is an ambispective study in which healthy patients without history of RIF and RM and with indication of egg donation cycle as ART treatment will be genotyped for KIR, HLA-C and HLA-F. Male partners and egg donors will also be studied for their HLA-C alleles. Patients would be assigned to donors, following routine clinical practice, without matching based on donor's HLA-C genotype. They would undergo SET and be followed up until delivery.

In addition to this prospective part, we will request access to data from patients who have equally undergone oocyte donation cycles at the clinic, who meet the inclusion criteria and who have been genotyped for KIR and HLA-C as a matter of routine practice.

Combinations of maternal KIR and HLA-C genotypes of the egg donor and fetus (based on the genotypes of the donor and male partner), as well as different HLA-F SNP genotypes of the recipients (form the prospective part of this proyect) will be correlated with reproductive outcomes. LBR will be the primary endpoint of the study. In addition, secondary endpoints such as embryo development, sustained implantation, progesterone leves, implantation failure and miscarriage rate will also be evaluated. Obstetrical complications such as preeclampsia, premature birth (<34 weeks) and low birth weight will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone or are undergoing their first egg donation cycle.
* Between 18 and 45 years of age.
* BMI between 19 and 25 kg/m2
* Signed written informed consent submitted.
* No history of RIF, defined as implantation failure after 4 consecutive blastocysts are transferred.
* No history of RM, defined as the presence of 2 or more clinical miscarriages.
* Normal blood pressure and viral serology.

Exclusion Criteria:

* Male partner diagnosed with severe male factor
* Patients who test positive for thrombophilic disorders (factor V Leiden, prothrombinG20210A mutation, positive antiphospholipid antibodies)
* Participation in a different study or clinical trial with a research drug or device in the last three months prior to recruitment.
* Known abnormal karyotype of subject or of her partner
* Any known clinically significant systemic disease
* Known inherited or acquired thrombophilia disease.
* Any known endocrine or metabolic abnormalities with the exception of controlled thyroid function disease.
* Severe psychiatric conditions.
* Patients with uterine factor/abnormalities (eg. myomas, polyps, adenomyosis, etc), that determines an unsatisfactory ultrasound for their ART.
* Patients with PCOS.
* Patients diagnosed with autoimmune diseases (eg. Systemic Lupus erythematosus, multiple sclerosis, rheumatoid arthritis).
* Patients with recent diagnosis (6 months) of chronic infectious disease (HPV, HBV, HCV, HIV, TBC).
* Patients with current treatment of immunosuppressant (eg. corticosteroids, monoclonal antibodies…).

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: The study population will consist of healthy patients with no history of RIF and RM which have undergone or are undergoing ART with oocyte donation and SET at IVI RMA Madrid, Valencia y Barcelona. Study subject candidates will be informed about the study once the inclusion criteria have been met. Data on reproductive outcomes, embryo development and perinatal and obstetric complications will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine if certain combinations of maternal KIR and oocyte donor HLA-C genotypes results in improved outcomes of live birth rate. | 36 months
  Principally, to establish whether patients of KIR AA and KIR Bx (2DS1-) genotypes show better outcomes when receiving oocytes from HLA-C1C1 donors than from donors with at least one HLA-C2 allele.

SECONDARY OUTCOMES:
To determine if certain combinations of maternal KIR and oocyte donor HLA-C genotypes results in improved outcomes of live birth rate taking into account the extra HLA-C2 alleles of the embryo. | 36 months
  To determine if certain combinations of maternal KIR and oocyte donor HLA-C genotypes results in improved outcomes of live birth rathe, in the same way as in the primary target, but taking into account the extra HLA-C2 alleles of the embryo with respect to the mother and the alternative division of the maternal genotypes into KIR AA, AB and BB.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Garcia Velasco, PhD, Principal Investigator — IVIRMA MADRID
Locations (1):
- Instituto Valenciano de Infertilidad, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No